CLINICAL TRIAL: NCT05403086
Title: Pragmatic Trial of Psilocybin Therapy in Palliative Care (PT2PC): A Multicenter Triple-blind Phase 2 Randomized Controlled Trial of Psilocybin Therapy for Demoralized Adults Near the End of Life
Brief Title: Pragmatic Trial of Psilocybin Therapy in Palliative Care
Acronym: PT2PC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Charles S. Grob, M.D. (Other)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Sponsor-Investigator, Charles S. Grob, M.D., Professor of Psychiatry and Behavioral Sciences, Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center
Organization: Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 21-008459
Record Dates: First submitted 2022-04-24; First posted 2022-06-03 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Demoralization
Keywords: Palliative Care; Serious Medical Illness; Life-threatening Condition; Advanced and Progressive Illness
MeSH Terms: interventions — Psilocybin; Hallucinogens; Ketamine

STUDY DESIGN:
Intervention Model Description: Parallel with optional Crossover for the control arm
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A Multicenter Triple-blind Phase 2 Randomized Controlled Trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Psilocybin (Experimental): A single moderate-to-high dose of oral psilocybin, plus 4-5 sessions of a brief, existential psychotherapy.
  Interventions: Drug: Psilocybin
- Ketamine (Active Comparator): A single low-to-moderate dose of oral liquid ketamine, plus 4-5 sessions of a brief, existential psychotherapy.
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Psilocybin — Psilocybin, [3-[2-(dimethylamino)ethyl]-1H-indol-4-yl] dihydrogen phosphate.
  Other Names: Hallucinogen
  Arms: Psilocybin
Drug: Ketamine — ketamine hydrochloride injection, for intravenous or intramuscular use, contains ketamine, a nonbarbiturate general anesthetic and has a molecular formula of C13H16ClNO•HCl and a molecular weight of 274.19. The chemical name for ketamine hydrochloride is (±)-2-(o-Chlorophenyl)-2-(methylamino)cyclohexanone hydrochloride.
  Other Names: Ketalar
  Arms: Ketamine

SUMMARY:
This multicenter, triple-blind, phase 2, randomized controlled trial will evaluate the efficacy and safety of psilocybin therapy compared to an active control in treating demoralization in adults near the end of life (≤2 years life expectancy).

DETAILED DESCRIPTION:
After providing written informed consent, participants deemed eligible for this trial will be randomized to a brief course of talk therapy plus 1 dose of oral psilocybin vs the same brief course of talk therapy plus 1 dose of oral ketamine (the active control). Participants' degree of demoralization and other clinical outcomes (e.g., depression, anxiety) will be assessed at 1, 2, and 5 weeks after the study drug administration. After completing the study, participants will have the option of being told which study drug they took (aka, "unblinded"); those who were randomized to the active control will be offered another brief course of talk therapy plus 1 dose of oral psilocybin, and the same sequence of outcome assessments.

ELIGIBILITY:
Inclusion Criteria:

General

* Provision of signed and dated informed consent form and the capacity to consent to research.
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Is currently a patient in a study-engaged clinical site
* Has a life-threatening illness and a life expectancy of ≤2 years
* Has moderate-to-severe demoralization
* Ability to take oral medication (capsules and liquid)

Exclusion Criteria:

General

* Known allergic or severe reactions to the non-psychoactive components of psilocybin capsules or liquid ketamine
* Treatment with another investigational drug or intervention within 1 month of signing Informed Consent Form (ICF)
* If deemed by clinical judgment of the study investigators to be unsafe for undergoing the intervention

Neurological

* Cognitive impairment sufficient to impede the ability to complete study tasks
* History of intracranial hemorrhage
* Recent embolic stroke
* Recent seizure
* Current intracranial mass
* Advanced stage of a neurologic disease that elevates risk for psychosis

Cardiovascular

* Uncontrolled hypertension
* Clinically significant cardiac disease

Respiratory

* Severe pulmonary disease
* Supplemental oxygen requirement

Gastrointestinal

* Current intractable nausea/vomiting/diarrhea
* Recent, clinically significant GI bleed
* Markedly abnormal liver function tests

Endocrine, Renal, and Reproductive

* Pregnancy or lactation
* Severe renal insufficiency
* Unstable insulin-dependent diabetes mellitus

Prohibited Medications

* Antipsychotics (with exceptions)
* Antidepressants (with exceptions)
* Dopamine agonists
* Drugs known to have adverse interactions with psilocybin or ketamine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-01-19 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in patient-reported Demoralization Scale-II.. | From Pre-dose V4 to ~14-days post drug (V8), and from Pre-dose (V4) to ~35-days post drug (V9), compared to active control.
  The DS-II is a validated, patient-reported outcome assessing demoralization with a 2-week recall period.

SECONDARY OUTCOMES:
i) Change in clinician-rated Clinical Global Impression (CGI) for Severity of demoralization. | From Enrollment (V1) to ~14-days (V8) and ~35-days (V9) post-drug for patients treated with psilocybin therapy vs active control.
  The CGI-I is a widely used and validated assessment of global clinical improvement. Possible scores range "0=Not assessed", "1=Very much improved", to "7=Very much worse." The CGI-I has been adapted here for assessing improvement in demoralization.
ii) Odds ratio of meeting criteria for demoralization on the clinician-rated Demoralization Interview Interview (DI). | From Enrollment (V1) to ~14-days (V8) and ~35-days (V9) post-drug for patients treated with psilocybin therapy vs active control.
  The CGI-I is a widely used and validated clinician-rated assessment of global clinical improvement. Possible scores range "0=Not assessed", "1=Very much improved", to "7=Very much worse." The CGI-I has been adapted here for assessing improvement in demoralization.
Change in depression symptoms | From Pre-dose V4 to ~14-days post drug (V8), and from Pre-dose V4 to ~35-days post drug (V9),
  A comparison to active control using the following measures: PHQ-9, GRID-HAM-D6.compared to active control
Change in anxiety symptoms, quality of life, and spiritual well-being | From Enrollment (V1) to ~14-days post drug (V8), and Enrollment (V1) to ~35-days post drug (V9)
  A comparison to active control, using the following measures: GAD-7, FACIT-Pal-14 FACIT-Sp-12.
Change in patient-reported pain | From Enrollment (V1) to ~14-days post drug (V8), and from Enrollment (V1) to ~35-days post drug (V9),
  A comparison to active control, using the Brief Pain Inventory-Short Form (BPI-SF).
Associations will be explored between change in Demoralization Scale-II and other measures pre-dose and 7 days post drug | From Pre-dose (V4) to 7-days post-drug.
  Associations will be explored between change in Demoralization Scale-II and 1) Credibility Expectancy Questionnaire (CrEQ), 2) Treatment Allocation Questionnaire, 3) Mystical Experience Questionnaire-30 (MEQ-30) and PEQ-4, 4) Challenging Experience Questionnaire (ChEQ), and 5) Change in Death Transcendence Scale-15 item (DTS-15)
DS-II and PHQ-9 comparison measures assessment | Throughout the study
  Change in DS-II and PHQ-9 will be compared to assess if there is a differential response to psilocybin therapy in this population.

CONTACTS AND LOCATIONS:
Overall Officials: Charles S. Grob, M.D., Principal Investigator — Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center
Locations (5):
- United States (5):
  - Marin Cancer Care, Greenbrae, California
  - University of California, Los Angeles, Los Angeles, California
  - University of San Francisco, San Francisco, California
  - Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center, Torrance, California
  - Sunstone Therapies, Rockville, Maryland

IPD SHARING:
Plan to Share IPD: Yes
Data from this study may be requested from other researchers 2 years after the completion of the primary endpoint by contacting the study sponsor.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will become available 2 years after completion of the primary endpoint.
Access Criteria: Data will be made available to qualified investigators who agree to the data sharing policies of the study.

REFERENCES:
- [Background] Gan LL, Gong S, Kissane DW. Mental state of demoralisation across diverse clinical settings: A systematic review, meta-analysis and proposal for its use as a 'specifier' in mental illness. Aust N Z J Psychiatry. 2022 Sep;56(9):1104-1129. doi: 10.1177/00048674211060746. Epub 2021 Dec 8. PMID 34879712
- [Background] Caruso R, Breitbart W. Mental health care in oncology. Contemporary perspective on the psychosocial burden of cancer and evidence-based interventions. Epidemiol Psychiatr Sci. 2020 Jan 9;29:e86. doi: 10.1017/S2045796019000866. PMID 31915100
- [Background] Reiche S, Hermle L, Gutwinski S, Jungaberle H, Gasser P, Majic T. Serotonergic hallucinogens in the treatment of anxiety and depression in patients suffering from a life-threatening disease: A systematic review. Prog Neuropsychopharmacol Biol Psychiatry. 2018 Feb 2;81:1-10. doi: 10.1016/j.pnpbp.2017.09.012. Epub 2017 Sep 22. PMID 28947181
- [Background] Ross S. Therapeutic use of classic psychedelics to treat cancer-related psychiatric distress. Int Rev Psychiatry. 2018 Aug;30(4):317-330. doi: 10.1080/09540261.2018.1482261. Epub 2018 Aug 13. PMID 30102082
- [Background] Robinson S, Kissane DW, Brooker J, Michael N, Fischer J, Franco M, Hempton C, Sulistio M, Pallant JF, Clarke DM, Burney S. Refinement and revalidation of the demoralization scale: The DS-II-internal validity. Cancer. 2016 Jul 15;122(14):2251-9. doi: 10.1002/cncr.30015. Epub 2016 May 12. PMID 27171617
- [Background] Robinson S, Kissane DW, Brooker J, Hempton C, Michael N, Fischer J, Franco M, Sulistio M, Clarke DM, Ozmen M, Burney S. Refinement and revalidation of the demoralization scale: The DS-II-external validity. Cancer. 2016 Jul 15;122(14):2260-7. doi: 10.1002/cncr.30012. Epub 2016 May 12. PMID 27171544
- [Background] Anderson BT, Danforth A, Daroff PR, Stauffer C, Ekman E, Agin-Liebes G, Trope A, Boden MT, Dilley PJ, Mitchell J, Woolley J. Psilocybin-assisted group therapy for demoralized older long-term AIDS survivor men: An open-label safety and feasibility pilot study. EClinicalMedicine. 2020 Sep 24;27:100538. doi: 10.1016/j.eclinm.2020.100538. eCollection 2020 Oct. PMID 33150319
- [Background] Grob CS, Danforth AL, Chopra GS, Hagerty M, McKay CR, Halberstadt AL, Greer GR. Pilot study of psilocybin treatment for anxiety in patients with advanced-stage cancer. Arch Gen Psychiatry. 2011 Jan;68(1):71-8. doi: 10.1001/archgenpsychiatry.2010.116. Epub 2010 Sep 6. PMID 20819978
- [Background] Ross S, Bossis A, Guss J, Agin-Liebes G, Malone T, Cohen B, Mennenga SE, Belser A, Kalliontzi K, Babb J, Su Z, Corby P, Schmidt BL. Rapid and sustained symptom reduction following psilocybin treatment for anxiety and depression in patients with life-threatening cancer: a randomized controlled trial. J Psychopharmacol. 2016 Dec;30(12):1165-1180. doi: 10.1177/0269881116675512. PMID 27909164
- [Background] Griffiths RR, Johnson MW, Carducci MA, Umbricht A, Richards WA, Richards BD, Cosimano MP, Klinedinst MA. Psilocybin produces substantial and sustained decreases in depression and anxiety in patients with life-threatening cancer: A randomized double-blind trial. J Psychopharmacol. 2016 Dec;30(12):1181-1197. doi: 10.1177/0269881116675513. PMID 27909165
- [Derived] Schipper S, Nigam K, Schmid Y, Piechotta V, Ljuslin M, Beaussant Y, Schwarzer G, Boehlke C. Psychedelic-assisted therapy for treating anxiety, depression, and existential distress in people with life-threatening diseases. Cochrane Database Syst Rev. 2024 Sep 12;9(9):CD015383. doi: 10.1002/14651858.CD015383.pub2. PMID 39260823